CLINICAL TRIAL: NCT06136611
Title: Preoperative Preradiotherapy TTFields (PORTRAIT)
Brief Title: Preoperative Preradiotherapy TTFields
Acronym: PORTRAIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other); Northern Care Alliance NHS Foundation Trust (Other); NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp221; 319109 (Other: IRAS)
Record Dates: First submitted 2023-01-09; First posted 2023-11-18 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Glioblastoma
Keywords: Neoadjuvant; Preoperative; Tumour Treating Fields
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: PORTRAIT is a cohort study including: 14 prospective patients for the experimental arm which assumes a TRUE toxicity rate of 20% (the study needs 13 patients and we allow 1 patient for replacement). This means that there is less than 10% chance that 4 or more patients will experience a toxicity defined as a complication. For the non-experimental arm, 28 prospective patients will be recruited.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optune (Experimental): Patients will apply TTFields (a treatment device referred to as Optune) before surgery and continue using this once the stitches are removed (approximately one to two weeks after surgery). Patients will wear the Optune application for 2 to 3 weeks before their standard-of-care (SoC) surgery and 3 to 4 weeks after the surgery (while awaiting their postoperative radiotherapy). Treatment with TTFields will be delivered through 4 transducer arrays with 9 insulated electrodes each placed on the shaved scalp and connected to a portable device set to generate 200-kHz electric fields within the brain.
  Interventions: Device: TTFields
- Non-Experimental Arm (No Intervention): Patients will follow the routine care pathway for glioblastoma and timings of the following will be determined by the clinical team.

INTERVENTIONS:
Device: TTFields — TTFields will be delivered through 4 transducer arrays with 9 insulated electrodes each placed on the shaved scalp and connected to a portable device set to generate 200-kHz electric fields within the brain.
  Arms: Optune

SUMMARY:
PreOperative PreRAdIotherapy Tumour Treating Fields (PORTRAIT) is a Phase I study that will test the safety and feasibility of Optune administered preoperatively and preradiotherapy in patients with a new radiological diagnosis of glioblastoma (GBM). Participants will be required to undergo additional MRI sequencing scans and provide blood, tear fluid and tissue samples over a maximum of 6 months. After the study patients will follow their standard treatment pathway.

DETAILED DESCRIPTION:
Glioblastoma is the most common primary malignant brain tumour in adults. Its outcomes are poor due to local disease progression in most patients. Current treatment includes surgery followed by chemotherapy and radiotherapy 4-6 weeks after surgery. In this time interval, some tumour cells do not receive any treatment. Furthermore, studies show that around half of all glioblastoma patients experience rapid early progression (REP) i.e. growth of the tumour in the time interval between surgery and postoperative chemotherapy/radiotherapy. REP is associated with a shorter survival and there are currently no effective treatments or preventative measures to address it.

Tumour Treating Fields (TTFields), also known as Optune, is a locally applied treatment modality that has contributed to a better survival outcome for glioblastoma patients when used after surgery and chemo-radiotherapy. We hypothesize that earlier treatment using the Optune device before the surgery and between the surgery and postoperative radiotherapy can prevent REP and improve patient outcome. In this phase 1 trial, PORTRAIT (PreOpeRaTive pRerAdIotherapy Ttfields), we will test the safety and feasibility of Optune treatment before surgery and before post-operative radiotherapy in a maximum of 14 patients. Participants will be required to undergo additional MRI sequencing scans and provide blood, tear fluid and tissue samples over a maximum of 6 months.

To maximise PORTRAIT's translational and clinically relevant components, a non-experimental arm (Non-EA) of 28 patients will allow comparisons of data collected from PORTRAIT patients with comparable Standard of Care (SoC) treated patients from the same time frame.

Participants will be invited to the research study if they are over the age of 35 and have a new radiological diagnosis of glioblastoma. All recruitment and treatment will be conducted at the Christie NHS Foundation Trust and Northern Care Alliance NHS Foundation Trust.

The study is funded by a research grant from Novocure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged >35 years (age range of more likely to suffer from an IDHwt WHO grade 4 astrocytoma)*
* Patient is male or female.
* Patient has a new radiological diagnosis of glioblastoma.
* Patient has a performance status judged by World Health Organisation, Eastern Cooperative Oncology Group [ECOG] score = 0-1.
* Patient has been reviewed by Neuro-oncology multidisciplinary team (MDT - neurosurgeon, clinical oncologist, radiologist and pathologist); MDT consensus that offering study entry is clinically appropriate and safe i.e. patient unlikely to come to harm (e.g. hydrocephalus) from delayed surgery and pre-operative Optune based on available clinical information and imaging.
* PI has confirmed at the first clinic visit that study entry is clinically appropriate and safe (e.g. lack of severe and debilitating symptoms of raised intracranial pressure).
* There is intention to treat the patient with surgical resection and postoperative adjuvant therapy as per current standard of care (40Gy/15 fr or 60Gy/30fr).
* Patient has adequate haematological and biochemical parameters for surgery and contrast agent administration (full blood count and coagulation profile deemed acceptable by clinical team, eGFR >30ml/min).
* Patient has mental capacity to consent for treatment.
* Patient is able and willing to give informed consent

Criteria specific to the experimental arm:

* Patient is able and willing to comply with study protocol requirements to continuously shave their head
* Patient is able and willing to comply with study protocol requirements to wear Optune equipment for the required duration.

Exclusion Criteria:

* Patients with uncontrolled seizures.
* Patients are due to undergo a planned biopsy procedure only.
* Patients have a suspicion of other tumour on CT body scan or known malignancy except non-melanoma skin cancer, completely resected or prostate cancer (with Prostate Specific Antigen of less than or equal to 0.1 ng/ml) within the past three years.
* Patients have contraindications to contrast-enhanced MRI scanning (e.g. claustrophobia, gadolinium allergy).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of Pre-Operative and Pre-Radiotherapy TTFields additional to the standard treatment of care (SoC) including adjuvant TTFields. | 18 months
  This endpoint will be tested by skin toxicity / wound complications.
  Toxicity is defined using CTCAE v5.0 and study related complications are defined as;
  * Skin toxicity grade 3 or higher
  * Wound closure or wound healing problems grade 2 or higher that are possibly related to TTFields treatment
To determine the incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of Pre-Operative and Pre-Radiotherapy TTFields additional to the standard treatment of care (SoC) including adjuvant TTFields. | 18 months
  This endpoint will be tested by alterations to the original date of surgery and the start of the postoperative radiotherapy;
  Study related complications will be defined as;
  * Change of surgery date due to symptoms related to the tumour that are possibly related to the TTFields treatment
  * Delay of start of the postoperative RT possibly related to the TTFields treatment (later than 6 weeks postoperative)

SECONDARY OUTCOMES:
Concordance between MRI based diagnosis of glioblastoma and definitive histological diagnosis | 18 months
  Evaluate the use of MRI to select glioblastoma patients for PORTRAIT without pathological confirmation.
REP: tumour volume difference between the post-operative MRI and pre-radiotherapy MRI. | 18 months
  Evaluate the effect of TTFields on REP - tumour growth between surgery and postoperative chemoradiotherapy, in patients with a new diagnosis of glioblastoma. A lower value represents a better outcome.
Registration of postoperative surgical complications | 18 months
  Postoperative surgical complications (e.g. haemorrhage, wound infection, delayed wound healing, seizures). Lower registrations represents a better outcome.
Registration of radiotherapy related complications | 18 months
  Radiotherapy related complications (e.g. radiation necrosis). Lower registrations represents a better outcome.
Steroid dose after TTFields | 18 months
  Steroid dose recorded after TTFields until the start of the postoperative RT. Lower (or absence of) dose represents a better outcome.
Progression free survival | 18 months
  Time period from the date of surgery to the date of the MRI scan demonstrating first progression as determined by the neuro-oncology MDT. A longer time period represents a better outcome.
Overall survival | 18 months
  Time period from the date of surgery to the date of death. A longer time period represents a better outcome.
Collection of liquid biopsies | 18 months
  Collection of blood and tear fluid samples at matched imaging timepoints.
Skin reactions | 18 month
  Skin reactions defined by CTCAE V5.0 - a rating scale of 1 to 5. 1 indicates minimal toxicity (skin irritation etc), 5 indicates death - or life threatening complications.

IPD SHARING:
Plan to Share IPD: Yes
Anonymised IPD relating to specified clinical outcomes may be shared upon request. A Sponsor approved Data Management Plan will detail the full sharing criteria and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Anonymised data will be made freely available following any temporary data embargos put in place by the funder or from researchers rights to the exclusive use of data (e.g. 6 months).
Access Criteria: Appropriate scientific justification, review by Principal Investigator and Trial Management Group, necessary legal contracts e.g. Data Access Agreements in place.